CLINICAL TRIAL: NCT04190511
Title: Characteristic and Modulation of Gut Microbiota on the Consequences of Pregnancy-based on the Maternal and Offspring Health Cohort
Brief Title: Characteristic and Modulation of Gut Microbiota on the Consequences of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Guanghui Li, Professor, MD, PhD, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-KY-015-01
Record Dates: First submitted 2019-11-27; First posted 2019-12-09 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Gestational Diabetes Mellitus; Medical Nutrition Therapy; Overweight/Obese; Gut Microbiota; Adverse Pregnancy Outcomes
MeSH Terms: conditions — Diabetes, Gestational; Overweight; Obesity | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prebiotic-containing dairy intervention group (Experimental)
  Interventions: Dietary Supplement: Prebiotic-containing dairy; Dietary Supplement: Dietary intervention
- Dietary intervention group (Active Comparator)
  Interventions: Dietary Supplement: Dietary intervention
- Conventional care group (No Intervention)

INTERVENTIONS:
Dietary Supplement: Prebiotic-containing dairy — The trained dietitian gives guidance on diet, exercise, and weight gain during pregnancy based on the Maternal Dietary Guidelines and Dietary Pagoda recommendations developed by the Chinese Institute of Maternal and Child Nutrition. On this basis, intervention was carried out using prebiotic-containing dairy products (200g/day).
  Arms: Prebiotic-containing dairy intervention group
Dietary Supplement: Dietary intervention — The trained dietitian gives guidance on diet, exercise, and weight gain during pregnancy based on the Maternal Dietary Guidelines and Dietary Pagoda recommendations developed by the Chinese Institute of Maternal and Child Nutrition.
  Arms: Dietary intervention group; Prebiotic-containing dairy intervention group

SUMMARY:
Since the incidence of maternal obesity and gestational diabetes mellitus (GDM) is on the rise globally, how to improve the intrauterine environment of the offspring and prevent obesity and metabolic diseases from the early life has become a medical research. Since 2012, journals such as Nature and Science have reported that intestinal micro-ecological environments composed of intestinal microbes and their interactions are involved in human body and energy metabolism, and a variety of metabolic diseases including obesity and type 2 diabetes mellitus (T2DM). The incidence is closely related. Although intestinal microbes have an important impact on human health, the research on intestinal microecology during pregnancy is still in its infancy. The current research is still unclear about the relationship between intestinal microecology and pregnancy outcomes and whether it can be a potential target for regulating maternal metabolism and fetal intrauterine environment. Therefore, this study aims to regulate overweight/obese pregnant women by using prebiotic-containing dairy products to explore the effects of interventions targeting intestinal microbes on glucose and lipid metabolism, insulin resistance and risk of GDM in overweight/obese pregnant women. In order to improve the intrauterine environment and reduce the risk of fetal diseases. It is of great significance and value to improve the quality of the birth population in China and to alleviate the medical economic burden caused by obesity and metabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 ~ 45 years
* single pregnancy
* enrollment week 8-12 + 6 weeks (based on the last menstrual period or B-ultrasound monitoring)
* BMI ≥ 25 kg / m2
* living in Beijing for at least 5 years

Exclusion Criteria:

* Taking antibiotics, probiotics or prebiotics
* smoking regularly
* drinking alcohol
* assisted fertility technology conception
* mental illness who were unable to answer questions correctly or were unwilling to conduct questionnaire surveys
* history of bariatric surgery
* not following dietary recommendations
* Lactose intolerance
* milk protein allergy
* pre-pregnancy hypertension, diabetes, Hyperlipidemia, hepatitis, nephritis, gastrointestinal diseases (chronic gastritis, enteritis, gastric ulcer and duodenal ulcer, etc.) and a history of infectious diseases (hepatitis, tuberculosis, etc.).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 375 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The incidence of gestational diabetes mellitus | Up to 28 weeks
  The diagnose of GDM based on the result of OGTT according to IADPSG criterion in 24 to 28 weeks. We will compare the incidence of GDM in these three groups.
Weight change during pregnancy | During pregnancy, an average of 38 weeks
  We asked pregnant woman to weigh their weight using the same weighing scale in the morning of the inspection day after urinating and tell the obstetrician to record. Compare the weight gain during pregnancy among three groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Obstetrics and Gynecology Hospital,Capital Medical University, Beijing, Chaoyang, China